CLINICAL TRIAL: NCT03513939
Title: A Safety, Tolerability and Efficacy Study of Sernova's Cell Pouch™ for Clinical Islet Transplantation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sernova Corp (Industry)
Collaborators: ICON plc (Industry); University of Chicago (Other); Breakthrough T1D (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROSVA201701
Record Dates: First submitted 2018-04-06; First posted 2018-05-02 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- T1D Cell Pouch Recipients (Experimental): Eligible Type 1 Diabetes Mellitus (T1D) subjects with hypoglycemia unawareness and a history of severe hypoglycemic episodes undergoing Sernova Cell Pouch intervention
  Interventions: Combination Product: Sernova Cell Pouch

INTERVENTIONS:
Combination Product: Sernova Cell Pouch — The Sernova Cell Pouch will be implanted against the rectus abdominis. The patient will receive either an 8-plug or 10-plug Cell Pouch configuration depending on Cohort assignment. A minimum of three weeks after Cell Pouch implantation, immunosuppression will be initiated and optimized for another 3 weeks. This will allow for proper vascularization of the Cell Pouch chambers and the patient to be stabilized on immunosuppression prior to islet transplantation. A mass of highly purified islets will be transplanted in the Cell Pouch.
  Patients who elect to retain the Cell Pouch after completion of the study will be asked to consent to long term safety follow-up, with data collected beyond the study scheduled visits every 3 months for up to 5 years until the last Cell Pouch explant (and then for a minimum of 3 months thereafter).

SUMMARY:
The Cell Pouch™ is a novel implantable device, that is transplanted with therapeutic cells such as insulin producing islets. This combination product is designed for the treatment of Type 1 Diabetes Mellitus (T1D) with hypoglycemia unawareness and a history of severe hypoglycemic episodes. Upon implantation, the Cell Pouch is designed to form a natural environment, rich in tissue and microvessels for the transplant and function of therapeutic cells. The Cell Pouch is designed as a scaffold made of non-degradable polymers, formed into small cylindrical chambers which, when implanted against the abdominal muscle, becomes incorporated with vascularized tissue to the circumference of removable plugs within as early as two weeks as demonstrated in preclinical studies. After the tissue incorporation, the plugs are removed, leaving fully formed tissue chambers with central void spaces for the transplantation of therapeutic cells including Islets of Langerhans (islets). Tissue integration within and around the Cell Pouch forms a natural environment, rich in microvessels that allows the transplanted islets to engraft, resulting in a functional biohybrid organ. It is believed this engraftment will enable long-term survival and function of transplanted islets. This study aims to demonstrate the safety and tolerability of islet transplantation into the Cell Pouch for the treatment of T1D in subjects with hypoglycemia unawareness and a history of severe hypoglycemic episodes. The study also aims to establish islet release criteria that accurately characterize the islet product and are predictive of clinical transplant outcomes into the Cell Pouch, which will be demonstrated through defined efficacy measures.

DETAILED DESCRIPTION:
The Sernova Cell Pouch is implanted against the abdominal musculature. A minimum of three weeks after Cell Pouch implantation, immunosuppression is initiated and optimized for another 3 weeks. This allows for vascularization of the Cell Pouch chambers and for the patient to be stabilized on immunosuppression prior to islet transplantation. A mass of highly purified islets will be transplanted in the Cell Pouch. The Cell Pouch will be assessed for safety and tolerability for up to five years (recently increased from 3 years) following the last transplant to Cell Pouch. Data for the primary and secondary endpoints will be summarized using descriptive statistics (such as counts and percentages).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 to 65 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Clinical history compatible with Type 1 Diabetes Mellitus (T1DM) with onset of disease at <40 years of age, insulin-dependence for ≥5 years at the time of consent, and a sum of patient age and insulin dependent diabetes duration of ≥28.
5. Absent stimulated c-peptide (<0.3 ng/mL) in response to a mixed meal tolerance test (MMTT; measured during the 4 hour test).
6. Involvement in intensive diabetes management defined as self-monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Such management must be under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least 3 clinical evaluations during the 12 months prior to study consent.
7. At least one episode of severe hypoglycemia in the 12 months prior to study consent.
8. Reduced awareness of hypoglycemia. More information about this criterion, including specific definitions of hypoglycemia unawareness, is in the protocol.

Exclusion Criteria:

1. Body mass index (BMI) >30 kg/m2
2. Insulin requirement >1.0 IU/kg/day
3. Glycated Haemoglobin (HbAlc) >13%.
4. Untreated proliferative diabetic retinopathy.
5. Blood Pressure: Systolic blood pressure (SBP) >160 mmHg or Diastolic Blood Pressure (DBP) >100 mmHg.
6. Measured glomerular filtration rate <70 mL/min/1.73m2 (More information about this criterion is in the protocol
7. Presence or history of macroalbuminuria (>300 mg/g creatinine).
8. Presence or history of panel-reactive anti-HLA antibodies >30%
9. For female subjects of child bearing potential: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. More information about this criterion is in the protocol.
10. Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
11. Patients with negative screen for Epstein Barr Virus by Immunoglobulin G (IgG) determination. More information about this criterion is in the protocol,
12. Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection within one year prior to study consent.
13. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
14. Active smoking, vaping or marijuana use or known active alcohol or substance abuse.
15. Baseline Hb below the lower limits of normal at the local laboratory for patients initially being enrolled into study.
16. Severe co-existing cardiac disease, characterized by any one of these conditions:

    * Recent myocardial infarction (within past 6 months).
    * Left ventricular ejection fraction <30%.
    * Uncontrolled coronary artery disease.
    * Known hypercoagulative state or
    * International Normalized Ratio > 1.8
17. Uncontrolled hyperlipidemia (fasting LDL cholesterol >130mg/dL and/or fasting triglycerides >200mg/dL).
18. Persistent elevation of liver function tests. More information on this criterion is in the protocol
19. Severe unremitting diarrhea, vomiting or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications (for example untreated celiac disease).
20. Untreated Graves' disease
21. Portal hypertension
22. Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≤ 5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
23. Treatment with any anti-diabetic medication other than insulin within 4 weeks of transplant, More information on this criterion is in the protocol
24. Use of any investigational agents within 4 weeks of consent
25. Administration of live attenuated vaccine(s) within 2 months of consent.
26. Any medical condition that, in the opinion of the study investigator, will interfere with safe participation in the trial.
27. Treatment with any immunosuppressive regimen at the time of consent.
28. A previous islet transplant.
29. A previous pancreas transplant. More information on this criterion is in the protocol
30. Known allergy or hypersensitivity to polymers More information on this criterion is in the protocol
31. Islets from non-heart beating donors will be excluded as well as from CDC high-risk donors.
32. Presence of colostomy/ileostomy, incisional hernia or other deformity of the abdominal wall precluding implantation of the Cell Pouch.
33. History of malignant hypertension or other conditions precluding general anesthesia.
34. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with prothrombin time (PT-INR) > 1.5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of the Cell Pouch following implantation, and islet transplantation, by evaluating the incidence and severity of adverse events (AEs) determined to be probable or highly probable to the Cell Pouch | 365 days ±14 days
  Safety will be assessed by evaluating the incidence and severity of adverse events (AEs) determined to be probable or highly probable to the Cell Pouch following initial Cell Pouch implantation, at the time of islet transplantation, and following islet transplantation, and throughout the study up to 365 days ±14 days post-islet transplantation

SECONDARY OUTCOMES:
Survival of endocrine tissue in the Cell Pouch (defined by positive staining of islets during histological analysis) | 90±5 days post-transplant for sentinel Cell Pouch
  Survival of endocrine tissue in the Cell Pouch (defined by positive staining of islets during histological analysis), as evaluated at day 90±5 days (post-removal of sentinel Mini Cell Pouch); or post-removal of Cell Pouches at any time during the study
Proportion of participants with a reduction in severe hypoglycemic events | From Day 0 to 90±5 ; Day 90±5 to Day 180±5; Day 180±5 to Day 365±14 following final Cell Pouch transplant and/or last transplant
  Proportion of participants, by cohort and in aggregate, with a reduction in severe hypoglycemic events following final Cell Pouch transplant and/or last islet transplant
Proportion of participants with a reduction in HbA1c >1mg% | From Day 0 to 90±5 ; Day 90±5 to Day 180±5; Day 180±5 to Day 365±14 following final Cell Pouch transplant and/or last transplant
  Proportion of participants, by cohort and in aggregate, with a reduction in HbA1c >1mg% following final Cell Pouch transplant and/or last islet transplant

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Witkowski, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No